CLINICAL TRIAL: NCT04537286
Title: A Prospective, Single-arm, Open-Label, Phase II Study of Nab-paclitaxel Plus Cisplatin Plus Carilizumab as First-line Treatment in Patients With Metastatic Triple-negative Breast Cancer
Brief Title: First-line Nab-paclitaxel Plus Cisplatin Plus Carilizumab in mTNBC Patients
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Biyun Wang, MD, Professor, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: YOUNGBC-11
Record Dates: First submitted 2020-08-29; First posted 2020-09-03 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — 130-nm albumin-bound paclitaxel; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- nab-paclitaxel plus cisplatin plus carilizumab (AP+PD-1) (Experimental): Nab-paclitaxel 125 mg/m2，ivgtt，d1, 8 Cisplatin 75 mg/m2，ivgtt，d1 Carilizumab 200mg, ivgtt，d1，q2w
  Interventions: Drug: nab-paclitaxel plus cisplatin plus carilizumab (AP+PD-1)

INTERVENTIONS:
Drug: nab-paclitaxel plus cisplatin plus carilizumab (AP+PD-1) — Nab-paclitaxel 125 mg/m2，ivgtt，d1, 8 Cisplatin 75 mg/m2，ivgtt，d1 Carilizumab 200mg, ivgtt，d1，q2w

SUMMARY:
To evaluate the efficacy and safety of nab-paclitaxel plus cisplatin plus carilizumab as first-line treatment in patients with metastatic triple-negative breast cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Female patients aged 18-70 years who had
2. Metastatic TNBC. ER, PgR, and HER2 status were determined locally by immunohistochemistry (IHC) of patient primary or metastatic tumor sections. Metastatic disease was confirmed by clinical, imaging, histological or cytological measures.
3. Patients were required to receive no previous chemotherapy or targeted therapy for metastatic triple-negative breast cancer.
4. Patients who had received adjuvant/neoadjuvant therapy were required an interval for at least 6 months after stop of chemotherapy before the enrollment.
5. At least one measurable lesion according to RECIST 1.1,
6. ECOG performance status ≤ 1
7. Life expectancy of more than 12 weeks
8. Adequate organ and bone marrow function.

Exclusion Criteria:

1. Patient of childbearing potential but unwilling to receive contraception.
2. Radiation therapy of axial bone within 4 weeks before enrollment.
3. Previous treatment with PD-1 antibody, PD-L1 antibody and CTLA-4 antibody.
4. Patients have active autoimmune diseases.
5. Patients who need systemic corticosteroids (> 10 mg prednisone/d) or other immunosuppressive drugs within 14 days before enrollment or during the study period.
6. Symptomatic central nervous system (CNS) disease (patients with asymptomatic treated CNS metastases were permitted)
7. Other malignant diseases within the past 5 years (patients with basal cell skin carcinoma and cervical carcinoma in situ were permitted)
8. Uncontrolled infection.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2020-08-25 (Actual); Primary Completion 2024-09-15 (Estimated); Study Completion 2024-10-15 (Estimated)

PRIMARY OUTCOMES:
PFS | 6 weeks
  Progression free survival
Adverse events | 6 weeks
  Number of participants with treatment-related adverse events as assessed by Common Terminology Criteria for Adverse Events version 4.0 (CTCAE v4.0)

CONTACTS AND LOCATIONS:
Overall Officials: Biyun Wang, Professor, Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No
Shared patient information is not allowed by study center.